CLINICAL TRIAL: NCT03378843
Title: Association Between Dietary Spermidine Intake and Mortality in the Population-based Bruneck Study
Brief Title: Spermidine Intake and All-cause Mortality
Status: Completed | Type: Observational
Sponsor: Medical University Innsbruck (Other)
Collaborators: Krankenhaus Bruneck (Other); University of Graz (Other); Paracelsus Medical University (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); King's College London (Other); Universitaet Innsbruck (Other)
Responsible Party: Principal Investigator, Stefan Kiechl, A.Univ.-Prof. Dr., Medical University Innsbruck
Other Study IDs: Bruneck_2017_Spermidine
Record Dates: First submitted 2017-12-14; First posted 2017-12-20 (Actual); Last update posted 2017-12-20 (Actual); Status verified 2017-12

CONDITIONS: Healthy Diet; Mortality
Keywords: Polyamine, cardiovascular disease, cancer
MeSH Terms: conditions — Cardiovascular Diseases; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Spermidine content of natural diet — The exposure consists in the long-term average dietary intake of the polyamine spermidine

SUMMARY:
This study seeks to test the potential association between spermidine content in diet and mortality in humans.

DETAILED DESCRIPTION:
This prospective community-based cohort study includes 829 participants aged 45-84 years, 49.9% of which are male. Diet is assessed by repeated dietician-administered validated food-frequency questionnaires (2540 assessments) in 1995, 2000, 2005, and 2010. Nutrient intakes including spermidine are calculated using USDA standard databases. Clinical events (all-cause mortality and cause-specific mortality) are recorded from 1995 to 2015.

The primary endpoint of all-cause mortality is related to the exposure of long-term average spermidine intake by Cox proportional hazards models with time-varying covariates. Additional analyses employ the Fine and Gray proportional subdistribution hazards model and flexible Royston-Parmar spline-based models. Comprehensive sensitivity analyses are performed to guard against potential biases associated with nutritional epidemiology.

ELIGIBILITY:
Inclusion Criteria:

Resident of Bruneck aged 40-79 years in 1990, age- and sex-stratified random sample.

Exclusion Criteria: None.

Ages: 45 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A random sample intended to represent the general population, recruited in 1990.
Sampling Method: Probability Sample
Enrollment: 829 (Actual)
Dates: Start 1995-10 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | 1995-2015
  Death due to any cause

SECONDARY OUTCOMES:
Cause-specific mortalities | 1995-2015
  Death due to cardiovascular disease, cancer, or other causes

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Kiechl, MD, Principal Investigator — Medical University of Innsbruck

IPD SHARING:
Plan to Share IPD: No
We do not plan to share individual participant data.

REFERENCES:
- [Background] Kiechl S, Lorenz E, Reindl M, Wiedermann CJ, Oberhollenzer F, Bonora E, Willeit J, Schwartz DA. Toll-like receptor 4 polymorphisms and atherogenesis. N Engl J Med. 2002 Jul 18;347(3):185-92. doi: 10.1056/NEJMoa012673. PMID 12124407
- [Background] Stegemann C, Pechlaner R, Willeit P, Langley SR, Mangino M, Mayr U, Menni C, Moayyeri A, Santer P, Rungger G, Spector TD, Willeit J, Kiechl S, Mayr M. Lipidomics profiling and risk of cardiovascular disease in the prospective population-based Bruneck study. Circulation. 2014 May 6;129(18):1821-31. doi: 10.1161/CIRCULATIONAHA.113.002500. Epub 2014 Mar 12. PMID 24622385
- [Background] Pechlaner R, Tsimikas S, Yin X, Willeit P, Baig F, Santer P, Oberhollenzer F, Egger G, Witztum JL, Alexander VJ, Willeit J, Kiechl S, Mayr M. Very-Low-Density Lipoprotein-Associated Apolipoproteins Predict Cardiovascular Events and Are Lowered by Inhibition of APOC-III. J Am Coll Cardiol. 2017 Feb 21;69(7):789-800. doi: 10.1016/j.jacc.2016.11.065. PMID 28209220
- [Derived] Kiechl S, Pechlaner R, Willeit P, Notdurfter M, Paulweber B, Willeit K, Werner P, Ruckenstuhl C, Iglseder B, Weger S, Mairhofer B, Gartner M, Kedenko L, Chmelikova M, Stekovic S, Stuppner H, Oberhollenzer F, Kroemer G, Mayr M, Eisenberg T, Tilg H, Madeo F, Willeit J. Higher spermidine intake is linked to lower mortality: a prospective population-based study. Am J Clin Nutr. 2018 Aug 1;108(2):371-380. doi: 10.1093/ajcn/nqy102. PMID 29955838